CLINICAL TRIAL: NCT01174849
Title: A Randomised Controlled Trial of Pneumococcal Conjugate Vaccines Synflorix and Prevenar13 in Sequence or Alone in High-risk Indigenous Infants (PREV-IX_COMBO): Immunogenicity, Carriage and Otitis Media Outcomes
Brief Title: Pneumococcal Vaccines Early and in Combination
Acronym: PREVIX_COMBO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 605810; ACTRN12610000544077 (Registry Identifier: Australia New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Otitis Media
Keywords: otitis media; pneumococcal vaccines; randomised controlled trial; high-risk children; indigenous; Australia
MeSH Terms: conditions — Otitis Media | interventions — PHiD-CV vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Synflorix (Active Comparator)
  Interventions: Drug: Synflorix
- Prevenar13 (Active Comparator)
  Interventions: Drug: Prevenar13
- COMBO (Experimental): COMBINATION SCHEDULE of comparator vaccine 1 and comparator vaccine 2 Synflorix at 1,2,4 months then Prevenar13 at 6 months.
  Interventions: Drug: COMBO

INTERVENTIONS:
Drug: Synflorix — The 10-valent vaccine contains 1 µg of purified capsular polysaccharide of pneumococcal serotypes 1, 5, 6B, 7F, 9V, 14, and 23F conjugated to protein D, 3 µg of serotype 4 conjugated to protein D, 3 µg of serotype 18C conjugated to tetanus toxoid and 3 µg of serotype 19F conjugated to diphtheria toxoid.
  Other Names: PHiD-CV
  Arms: Synflorix
Drug: Prevenar13 — The vaccine is a ready to use homogeneous white suspension for intramuscular injection, supplied as a pre-filled syringe.
  Active ingredients
  Each 0.5 mL dose contains:
  2.2 μg of pneumococcal purified capsular polysaccharides for serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F and 23F 4.4 μg of pneumococcal purified capsular polysaccharides for serotype 6B. Each serotype is individually conjugated to non-toxic diphtheria CRM197 protein and adsorbed on aluminium phosphate (0.565 mg). CRM197 is a nontoxic variant of diphtheria toxin isolated from cultures of Corynebacterium diphtheriae strain C7 (β197) grown in a casamino acids and yeast extract-based medium.
  Other Names: PCV13
  Arms: Prevenar13
Drug: COMBO — COMBINATION SCHEDULE of vaccine 1 and vaccine 2: Synflorix (PHiD-CV) at 1,2,4 months then Prevenar13 (PCV13) at 6 months of age.
  Other Names: Combination schedule
  Arms: COMBO

SUMMARY:
The purpose of this study is to determine whether an early schedule of a combination of three doses of PHiD-CV and one dose of PCV13, is superior to three doses of either PCV13 or PHiD-CV.

DETAILED DESCRIPTION:
Aboriginal children in the Northern Territory (NT) have high rates of otitis media caused by non-capsular H. influenzae (NCHi) and pneumococci. Pneumococcal conjugate vaccine has effectively reduced disease caused by the 7 serotypes. Rates of non-vaccine serotype otitis media (OM), particularly 19A is increasing, and NCHi continues to be a major pathogen in perforations. Parallels with pneumonia are highly probable in this population. Vaccines with expanded and early age protection are needed.

In early 2009 GSK's pneumococcal H. influenzae protein D conjugate vaccine (PHiD-CV) was licensed in Australia. Compared to the current vaccine, 7PCV, this vaccine offers protection from pneumococcal serotypes 1, 5, 7F as well as NCHi (which is a primary pathogen of OM, and possibly pneumonia). However by 2010, a new generation of Wyeth's 7PCV, PCV13 will also be licensed in Australia. Compared to PHiD-CV this vaccine offers protection from additional serotypes 3, 6A and 19A, however it does not offer protection from NCHi infection. There is no empirical evidence to suggest that either vaccine will have superior clinical efficacy for otitis media or pneumonia in high-risk children. The novel combination strategy proposed for this trial has the potential to provide the best of both vaccines.

ELIGIBILITY:
Inclusion Criteria:

Indigenous infants

* 4 to 6 weeks of age
* Living in remote communities that have provided signed Expressions of Interest in participating in PREV-IX_COMBO trial
* Intend to remain in their community until their baby is 7 months of age
* Eligible for routine vaccinations.

Exclusion Criteria:

* Prior adverse reaction to pneumococcal conjugate vaccines according to Australian Immunization Handbook.
* Gestational age < 32 weeks

Ages: 28 Days to 38 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 425 (Actual)
Dates: Start 2011-08; Primary Completion 2017-09-21 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 7 months of age
  At 7 months of age, the overall and serotype specific (particularly serotype 19A and HiD) a IgG Geometric Mean Concentration (GMC) b proportion of children with IgG GMC above threshold (0.35 microg/mL)

SECONDARY OUTCOMES:
nasopharyngeal carriage | 7 months of age
  At 7 months of age, the proportion of children with any carriage of serotype 19A pneumococci
nasopharyngeal carriage | 7 months of age
  At 7 months of age, the proportion of children with any carriage of non-capsular H. influenzae.
otitis media | 7 months of age
  At 7 months of age, the proportion of children with any otitis media.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Leach, PhD, Principal Investigator — Menzies School of Health Research
Locations (1):
- Menzies School of Health Research, Darwin, Northern Territory, Australia

REFERENCES:
- [Background] Morris PS, Leach AJ, Silberberg P, Mellon G, Wilson C, Hamilton E, Beissbarth J. Otitis media in young Aboriginal children from remote communities in Northern and Central Australia: a cross-sectional survey. BMC Pediatr. 2005 Jul 20;5:27. doi: 10.1186/1471-2431-5-27. PMID 16033643
- [Background] Leach AJ, Morris PS. The burden and outcome of respiratory tract infection in Australian and aboriginal children. Pediatr Infect Dis J. 2007 Oct;26(10 Suppl):S4-7. doi: 10.1097/INF.0b013e318154b238. PMID 18049380
- [Background] Leach AJ, Morris PS, Mathews JD; Chronic Otitis Media Intervention Trial - One (COMIT1) group. Compared to placebo, long-term antibiotics resolve otitis media with effusion (OME) and prevent acute otitis media with perforation (AOMwiP) in a high-risk population: a randomized controlled trial. BMC Pediatr. 2008 Jun 2;8:23. doi: 10.1186/1471-2431-8-23. PMID 18513453
- [Background] Leach AJ, Morris PS, Mackenzie G, McDonnell J, Balloch A, Carapetis J, Tang M. Immunogenicity for 16 serotypes of a unique schedule of pneumococcal vaccines in a high-risk population. Vaccine. 2008 Jul 23;26(31):3885-91. doi: 10.1016/j.vaccine.2008.05.012. Epub 2008 May 27. PMID 18562052
- [Background] Leach AJ, Morris PS, McCallum GB, Wilson CA, Stubbs L, Beissbarth J, Jacups S, Hare K, Smith-Vaughan HC. Emerging pneumococcal carriage serotypes in a high-risk population receiving universal 7-valent pneumococcal conjugate vaccine and 23-valent polysaccharide vaccine since 2001. BMC Infect Dis. 2009 Aug 4;9:121. doi: 10.1186/1471-2334-9-121. PMID 19650933
- [Background] Mackenzie GA, Carapetis JR, Leach AJ, Morris PS. Pneumococcal vaccination and otitis media in Australian Aboriginal infants: comparison of two birth cohorts before and after introduction of vaccination. BMC Pediatr. 2009 Feb 19;9:14. doi: 10.1186/1471-2431-9-14. PMID 19228431
- [Background] Leach AJ, Boswell JB, Asche V, Nienhuys TG, Mathews JD. Bacterial colonization of the nasopharynx predicts very early onset and persistence of otitis media in Australian aboriginal infants. Pediatr Infect Dis J. 1994 Nov;13(11):983-9. doi: 10.1097/00006454-199411000-00009. PMID 7845752
- [Background] Smith-Vaughan H, Byun R, Nadkarni M, Jacques NA, Hunter N, Halpin S, Morris PS, Leach AJ. Measuring nasal bacterial load and its association with otitis media. BMC Ear Nose Throat Disord. 2006 May 10;6:10. doi: 10.1186/1472-6815-6-10. PMID 16686940
- [Background] Hare KM, Morris P, Smith-Vaughan H, Leach AJ. Random colony selection versus colony morphology for detection of multiple pneumococcal serotypes in nasopharyngeal swabs. Pediatr Infect Dis J. 2008 Feb;27(2):178-80. doi: 10.1097/INF.0b013e31815bb6c5. PMID 18174871
- [Background] Prymula R, Peeters P, Chrobok V, Kriz P, Novakova E, Kaliskova E, Kohl I, Lommel P, Poolman J, Prieels JP, Schuerman L. Pneumococcal capsular polysaccharides conjugated to protein D for prevention of acute otitis media caused by both Streptococcus pneumoniae and non-typable Haemophilus influenzae: a randomised double-blind efficacy study. Lancet. 2006 Mar 4;367(9512):740-8. doi: 10.1016/S0140-6736(06)68304-9. PMID 16517274
- [Background] Roche PW, Krause V, Cook H, Barralet J, Coleman D, Sweeny A, Fielding J, Giele C, Gilmour R, Holland R, Kampen R; Enhanced Invasive Pneumococcal Disease Surveillance Working Group; Brown M, Gilbert L, Hogg G, Murphy D; Pneumococcal Working Party of the Communicable Diseases Network Australia. Invasive pneumococcal disease in Australia, 2006. Commun Dis Intell Q Rep. 2008 Mar;32(1):18-30. doi: 10.33321/cdi.2008.32.3. PMID 18522302
- [Derived] Leach AJ, Wilson N, Arrowsmith B, Beissbarth J, Mulholland K, Santosham M, Torzillo PJ, McIntyre P, Smith-Vaughan H, Skull SA, Oguoma VM, Chatfield MD, Lehmann D, Brennan-Jones CG, Binks MJ, Licciardi PV, Andrews RM, Snelling T, Krause V, Carapetis J, Chang AB, Morris PS. Hearing loss in Australian First Nations children at 6-monthly assessments from age 12 to 36 months: Secondary outcomes from randomised controlled trials of novel pneumococcal conjugate vaccine schedules. PLoS Med. 2024 Jun 3;21(6):e1004375. doi: 10.1371/journal.pmed.1004375. eCollection 2024 Jun. PMID 38829821
- [Derived] Leach AJ, Wilson N, Arrowsmith B, Beissbarth J, Mulholland EK, Santosham M, Torzillo PJ, McIntyre P, Smith-Vaughan H, Chatfield MD, Lehmann D, Binks M, Chang AB, Carapetis J, Krause V, Andrews R, Snelling T, Skull SA, Licciardi PV, Oguoma VM, Morris PS. Immunogenicity, otitis media, hearing impairment, and nasopharyngeal carriage 6-months after 13-valent or ten-valent booster pneumococcal conjugate vaccines, stratified by mixed priming schedules: PREVIX_COMBO and PREVIX_BOOST randomised controlled trials. Lancet Infect Dis. 2022 Sep;22(9):1374-1387. doi: 10.1016/S1473-3099(22)00272-9. Epub 2022 Jun 27. PMID 35772449
- [Derived] Leach AJ, Mulholland EK, Santosham M, Torzillo PJ, McIntyre P, Smith-Vaughan H, Wilson N, Arrowsmith B, Beissbarth J, Chatfield MD, Oguoma VM, Morris PS. Otitis media outcomes of a combined 10-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine and 13-valent pneumococcal conjugate vaccine schedule at 1-2-4-6 months: PREVIX_COMBO, a 3-arm randomised controlled trial. BMC Pediatr. 2021 Mar 8;21(1):117. doi: 10.1186/s12887-021-02552-z. PMID 33685411
- [Derived] Leach AJ, Mulholland EK, Santosham M, Torzillo PJ, Brown NJ, McIntyre P, Smith-Vaughan H, Skull S, Balloch A, Andrews R, Carapetis J, McDonnell J, Krause V, Morris PS. Pneumococcal conjugate vaccines PREVenar13 and SynflorIX in sequence or alone in high-risk Indigenous infants (PREV-IX_COMBO): protocol of a randomised controlled trial. BMJ Open. 2015 Jan 16;5(1):e007247. doi: 10.1136/bmjopen-2014-007247. PMID 25596202